CLINICAL TRIAL: NCT03372759
Title: Tilt of the Intraocular Lens in Patients Undergoing Combined Phacoemulsification and Vitrectomy With Airtamponade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of the department of Ophthalmology, principal investigator, Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: til
Record Dates: First submitted 2016-11-08; First posted 2017-12-14 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Epiretinal Membrane
MeSH Terms: conditions — Epiretinal Membrane | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- study group air (Active Comparator): airtamponade
  Interventions: Procedure: airtamponade
- study group saline (Sham Comparator): saline
  Interventions: Procedure: saline

INTERVENTIONS:
Procedure: airtamponade — airtamponade is applicated in the study group air
  Arms: study group air
Procedure: saline — saline is left in the study Group saline
  Arms: study group saline

SUMMARY:
Vitrectomy with membrane peeling has developed to be the gold-standard in treatment of epiretinal membranes. Due to the possibility of vitrectomy induced cataract, in many ophthalmic surgical centers it has become usual to indicate combined phacoemulsification and vitrectomy in case of existing cataract.

Epiretinal membranes (ERM) and pseudomaculaforamen are disorders involving the posterior pole of the eyeball with consecutive vision loss. ERM can be well visualized with spectral domain optical coherence tomography (SD-OCT). Different study groups showed that even intraoperative use of SD-OCT is possible.

DETAILED DESCRIPTION:
The aim of the study is to document tilt of the intraocular lens in combined phacoemulsification and vitrectomy by photography of purkinjereflexes. During vitrectomy tamonade with air or saline are regarded as equal in substituting the removed vitreous. In case of airtamponade, air will be resolved within several days. As airtamponade induces more anterior movement of the implanted intraocular lens in the superior parts of the lens, tilt can result. Saline doesn´t have any influence on the intraocular lens.

ELIGIBILITY:
Inclusion Criteria:

* patients sheduled for combined phakoemulsification and 23G pars plana vitrectomy
* Minimum Age of 21 years
* written informed consent

Exclusion Criteria:

* none

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-12; Primary Completion 2017-05 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
postoperative tilt of the IOL is measured with purkinjemetry | 3 months
  airtamponade has the potential to leave postoperative tilt of the IOL

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- VIROS - Vienna Institute for Research in Ocular Surgers - Departement of Opthalmology - Hanusch Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided